CLINICAL TRIAL: NCT03100669
Title: Implementing a Postoperative MIRP (Minimally Invasive Repair of Pectus) Program: Short and Long-term Evaluation of Pain, Nausea, Sleep, and Rehabilitation Via Tele-monitoring
Brief Title: Implementing a Postoperative MIRP (Minimally Invasive Repair of Pectus) Program Via Tele-monitoring
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, Davina Wildemeersch, Resident anesthesiology, University Hospital, Antwerp
Other Study IDs: 17/08/082
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain; Postoperative Nausea
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pectus surgery: Single arm study: patient undergoing pectus repair surgery
  Interventions: Procedure: Pectus surgery

INTERVENTIONS:
Procedure: Pectus surgery — Patients undergoing surgical repair of pectus excavatum or carinatum

SUMMARY:
MIRP (Minimally Invasive Repair of Pectus) as surgical correction of pectus excavatum or carinatum is performed to achieve physiological, cosmetic, and psychological benefits for the patient. Surgery is often associated with severe postoperative pain. In this study the researchers want to registrate pain, sleep, nausea/vomiting, and daily activities in short and long term follow up.

DETAILED DESCRIPTION:
In order to provide pain patients with an individualized approach to their pain problem after MIRP we developed an electronic medical record coupled to a set of telemetric medical-grade devices. Appi@Home (Antwerp Personalized Pain Initiative) supports an innovative approach to (sub)acute conditions by offering a platform for continuous follow-up. Patients are provided with a toolbox and an app that continuously collects objective outcome data (i.e. pain intensity, sleep quality, physical activity). The integrated system allows the care givers to respond very quickly to changing clinical conditions of the patient, making a very adaptive and individualized follow-up possible for these patients. In addition, the patient becomes an active participant in the global therapeutic approach.

Patients receive the toolbox two week prior to surgery with access to the internet platform for questionnaires fill-in procedure. Up to ten week after surgery pain intensity, sleep quality and physical activity will be monitored subjectively by a scoring table (0-10, 0 no pain-bad sleeping quality-no activity, 10 maximum of pain-excellent sleeping quality- a lot of activity) and objectively by blood pressure device, oxygen saturation monitoring, activity tracker and sleep registration tool.

ELIGIBILITY:
Inclusion Criteria:

* elective pectus repair
* signed informed consent

Exclusion Criteria:

* chronic opioid use (> 3 months)
* history of ongoing psychiatric disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients planned for elective pectus surgery are asked for study inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Pain | 10 weeks after surgery
  pain registration via numeric rating scale during hospitalization up to 10 weeks after surgery

SECONDARY OUTCOMES:
Sleep | 2 weeks before up to 10 weeks after surgery
  hours of sleep up to 10 weeks after surgery
Daily activity | 2 weeks before up to 10 weeks after surgery
  daily activity via scale (0: no activity and 10 maximum of activities) and activity tracker device during hospitalization up to 10 weeks after surgery
Nausea | From day of surgery until hospital discharge (approximately 7 days)
  registration of nausea and vomiting by questionnaire during hospitalization period
Mobility | From day of surgery until hospital discharge (approximately 7 days)
  Daily mobility assessment by attending physiotherapist via scale (1: exercises in bed, 2: exercises while sitting, 3: exercises while standing, 4: exercises while walking) during hospitalization

OTHER OUTCOMES:
Rosenberg self-esteem questionnaire | Allowed period for fill in: from two weeks before planned surgery until day before planned surgery
  Preoperative evaluation of self-esteem by the Rosenberg self-esteem questionnaire, via a patient specific online platform
Hospital anxiety and depression scale (HAD) | Allowed period for fill in: from two weeks before planned surgery until day before planned surgery
  Preoperative evaluation of anxiety and depression by the HAD questionnaire, via a patient specific online platform
State-Trait anxiety Inventory (STAI) | Allowed period for fill in: from two weeks before planned surgery until day before planned surgery
  Preoperative evaluation of state and trait characteristics by the STAI questionnaire, via a patient specific online platform
Multidisciplinary Pain Inventory (MPI) | Allowed period for fill in: first two weeks after hospital discharge
  Postoperative evaluation of pain severity and interference by the MPI questionnaire, via a patient specific online platform
Coping Pain Questionnaire (CPQ) | Allowed period for fill in: first two weeks after hospital discharge
  Postoperative evaluation of coping strategy (active, passive, self-efficacy) by the CPQ questionnaire, via a patient specific online platform

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wildemeersch D, D'Hondt M, Bernaerts L, Mertens P, Saldien V, Hendriks JM, Walcarius AS, Sterkens L, Hans GH. Implementation of an Enhanced Recovery Pathway for Minimally Invasive Pectus Surgery: A Population-Based Cohort Study Evaluating Short- and Long-Term Outcomes Using eHealth Technology. JMIR Perioper Med. 2018 Oct 12;1(2):e10996. doi: 10.2196/10996. PMID 33401363
- [Derived] Wildemeersch D, Bernaerts L, D'Hondt M, Hans G. Preliminary Evaluation of a Web-Based Psychological Screening Tool in Adolescents Undergoing Minimally Invasive Pectus Surgery: Single-Center Observational Cohort Study. JMIR Ment Health. 2018 May 31;5(2):e45. doi: 10.2196/mental.9806. PMID 29853436